CLINICAL TRIAL: NCT05363709
Title: A Phase 2 Study to Assess the Effect of BALSTILIMAB (AGEN2034) on Viral Clearance in HPV-positive Oropharyngeal Cancer Patients With Persistent HPV Detection in Plasma cfDNA After Definitive Therapy
Brief Title: BALSTILIMAB on Viral Clearance in HPV+ Oropharyngeal Cancer Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Agenus Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-1077; NCI-2022-03805 (Other: NCI-CTRP-Clinical Trial Reporting Registry)
Record Dates: First submitted 2022-04-26; First posted 2022-05-06 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: HPV; Oropharyngeal Cancer
MeSH Terms: conditions — Oropharyngeal Neoplasms | interventions — balstilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Balstilimab (Experimental): Participants will receive Balstilimab by vein over about 30 minutes on Days 1 and 15 of each cycle (every 2 weeks)
  Interventions: Drug: Balstilimab

INTERVENTIONS:
Drug: Balstilimab — Given by Vein (IV)
  Other Names: Balstilimab IB

SUMMARY:
This study aims to leverage this unique property of HPV+ OPC to detect possible minimal residual disease represented by persistent viral detection after the completion of definitive treatment. The study will offer adjuvant immune therapy to patients with persistent viral detection and evaluate the clearance of viral load. It will evaluate the rate of viral clearance with immune therapy and establish the link between viral clearance and long-term disease control.

DETAILED DESCRIPTION:
Objectives:

Primary Objective:

To assess whether anti-PD1 will lead to the clearance of the virus in the plasma cfDNA in HPV+ OPC patients with persistent cfDNA HPV following definitive therapy

Secondary Objectives:

* One-year recurrence-free survival (1-yr RFS),
* 2-year RFS (2-yr RFS),
* Overall survival (2-yr OS),
* Safety and tolerability
* Compliance
* Quality of life (EORTC C30 will be utilized)

Correlative/Exploratory Objectives:

* Time to viral clearance in the oral rinse and plasma cfDNA with anti-PD1 treatment
* The concordance between plasma HPV and oral rinse HPV at diagnosis, post-definitive treatment and during adjuvant treatment
* The correlation between tumor mutations and persistence of HPV in oral rinse/cfDNA.
* The correlation between recurrence site (loco-regional vs. distant metastasis) and oral rinse vs. plasma HPV detection

ELIGIBILITY:
Inclusion Criteria:

Subject must meet all of the following applicable inclusion criteria to participate in this study:

1. Written informed consent and HIPAA authorization for release of personal health information prior to registration. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
2. Histologically or cytologically confirmed squamous cell carcinoma from oropharynx. note: patients with a clinical diagnosis of oropharyngeal cancer, awaiting a biopsy is eligible to consent for prescreening.
3. Stage I-III per AJCC 8th edition
4. Positive p16 immunohistochemistry or HPV testing, or p16/HPV status unknown with patients having a less than 10 pack-year smoking history
5. Age ≥ 18 years at the time of consent.
6. Eastern Cooperative Oncology Group (ECOG) performance status 0-1 for patients who receive treatment
7. Persistent detection of cfDNA HPV (≥ 16 copies/mL) in the absence of clinically evident disease at 3, 6, or 9 months following definitive treatment (surgery, systemic therapy, and/or radiation therapy).
8. Patients must have adequate hematologic, coagulation, hepatic, and renal function for anti-PD1 treatment. this includes:

   * ANC >/= 1,500/mm3
   * platelet count >/=100,000/mm3
   * HgB ≥ 9 g/dL (may be with transfusion)
   * Creatinine ≤ 1.5x ULN or creatinine clearance (measured via 24-hour urine collection) ≥40 mL/minute (that is, if serum creatinine is >1.5 times the ULN, a 24-hour urine collection to calculate creatinine clearance must be performed).
   * Total Serum Bilirubin ≤ 1.5 x ULN (Patients with known Gilbert Syndrome, a total bilirubin ≤ 3.0 x ULN, with direct bilirubin ≤ 1.5 x ULN)
   * SGOT, SGPT ≤ 3 X ULN
   * SGOT, SGPT ≤ 5 X ULN
9. Females of childbearing potential must not be breast feeding and must have a negative pregnancy test during screening and 7 days prior to initiation of study treatment. The patient must agree to use adequate contraception. Note: women will be considered post-menopausal if they have been amenorrheic for the past 12 months without an alternative medical cause. The following agespecific requirements must also apply: women < 50 years old: they would be considered postmenopausal if they have been amenorrheic for the past 12 months or more following cessation of exogenous hormonal treatments. The levels of luteinizing hormone (LH) and follicle-stimulating hormone (FSH) must also be in the post-menopausal range (as per the institution). Women ≥ 50 years old: they would be considered post-menopausal if they have been amenorrheic for the past 12 months or more following cessation of all exogenous hormonal treatments, or have had radiation-induced oophorectomy with the last menses > 1 year ago, or have had chemotherapyinduced menopause with >1 year interval since last menses, or have had surgical sterilization by either bilateral oophorectomy or hysterectomy.
10. Non-sterilized males who are sexually active with a female partner of childbearing potential must use adequate contraception for the duration of the study.

Exclusion Criteria:

Subjects should not enter the study if any of the following exclusion criteria are fulfilled:

1. Prior treatment history with anti-PD-1 or anti-PD-L1 therapies are not allowed.
2. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses, which in the investigator's opinion makes it undesirable for the subject to participate in the trial or which would jeopardize compliance with the protocol, or active and uncontrolled infection including hepatitis B, hepatitis C and human immunodeficiency virus (HIV).

   Screening for chronic conditions is not required.
3. Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirement.
4. Active rheumatological or autoimmune conditions requiring systemic treatment, such as steroids.
5. Any evidence of current interstitial lung disease (ILD) or pneumonitis or a prior history of ILD or noninfectious pneumonitis requiring high-dose glucocorticoids.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-10-18 (Actual); Primary Completion 2028-02-15 (Estimated); Study Completion 2028-02-15 (Estimated)

PRIMARY OUTCOMES:
To establish the Overall survival. | through study completion, an average of 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Luana Guimaraes de Sousa, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org